CLINICAL TRIAL: NCT01069224
Title: Analysis of Proinflammatory Factors in the Synovial Fluid In Patients With Rotator Cuff Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Maman Eran MD, Tel Aviv Medical Center
Other Study IDs: MozesG
Record Dates: First submitted 2010-02-09; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Rotator Cuff Disease
Keywords: rotator cuff; synovial fluid; proinflammatory cytokines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid lavages will be collected at the time of arthroscopic RC reconstruction or other shoulder arthroscopy that will be performed for therapeutic goals (instability repair, SLAP lesion).

GROUPS / COHORTS (2):
- RC tear: This study will include a consecutive series of patients who met the study inclusion criteria. Study group patients will be diagnosed RC tear on clinical examination and imaging findings (US and MRI) that will be verified at arthroscopy in order to complete the enrollment.
- Control group: Control group will include patients suffering from shoulder instability that scheduled for elective surgical repair.

SUMMARY:
Role of proinflammatory factors in Patients with Rotator Cuff Disease

Objective:

To measure the levels of various cytokines and metalloproteases in patients with rotator cuff disease, and control group and to determine the correlations among them.

DETAILED DESCRIPTION:
We hypothesize that cytokines and MMP's level will be significantly higher in patients with RC pathology than in control group and will be related to the time frame since injury (i.e. - higher levels as close to the injury). In addition we will examine possible relation of those levels to the pain curve by using Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and accept the trial procedures and to sign an informed consent form in accordance with national legislation.
2. Patients between age 18-65 scheduled for a surgery in a Shoulder unit
3. Patients suffering from Rotator Cuff Disease
4. Patients suffering from any noninflammatory shoulder condition which requires surgical intervention

Exclusion Criteria:

1. Revision rotator cuff repair
2. Recurrent shoulder surgery
3. Psychiatric illness
4. Inflammatory condition.
5. Current use of anti-inflammatory drugs.
6. Previous or current shoulder infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a consecutive series of patients who met the study inclusion criteria. Study group patients will be diagnosed RC tear on clinical examination and imaging findings (US and MRI) that will be verified at arthroscopy in order to complete the enrollment.
  Control group will include patients suffering from shoulder instability that scheduled for elective surgical repair.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
cytokines and MMP's levels in patients with RC pathology and in control group | 12 month

SECONDARY OUTCOMES:
Levels of pain curve by using Visual Analogue Scale | 12 month